CLINICAL TRIAL: NCT01072760
Title: Kirschner Wire and Pull-out Wire Fixation for the Treatment of Bony Mallet Finger
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Second Hospital of Qinhuangdao (Other)
Responsible Party: Xu Zhang, The Second Hospital of Qinhuangdao
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: QHD201002; QHD20010201 (Other: The second hospital of Qinhuangdao)
Record Dates: First submitted 2010-02-12; First posted 2010-02-22 (Estimated); Last update posted 2010-02-22 (Estimated); Status verified 2010-02

CONDITIONS: Bony Mallet Finger
Keywords: Mallet finger; extensor tendon; Kirschner wire; Fracture Fixation
MeSH Terms: interventions — Bone Wires

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- K wire (Experimental)
  Interventions: Procedure: K wire

INTERVENTIONS:
Procedure: K wire — Mallet finger treatment
  Other Names: stainless steel wire

SUMMARY:
The objective of this report is to describe a new surgical technique for the treatment of bony mallet finger which involves the application of both Kirschner wire and pull-out wire fixation. It is believed to decrease the risk of the complications.

DETAILED DESCRIPTION:
From May 2003 to December 2008, we used Kirschner wire and pull-out wire fixation to carry out 54 closed bony mallet finger in 54 patients. The bony mallet finger was applicated both Kirschner wire and pull-out wire fixation.

ELIGIBILITY:
Inclusion Criteria:

1. bony mallet finger;
2. patient had failed trials of nonsurgical treatment;
3. fracture involving more than 1/3 of the joint surface;
4. fragment displacement or subluxation of the DIP joint.

Exclusion Criteria:

1. tendinous mallet finger;
2. success of nonsurgical treatment;
3. comminuted fracture;
4. fracture involving at or less than 1/3 of the joint surface which could be successfully replaced with nonsurgical treatment.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2003-05; Primary Completion 2008-12 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
The digits were assessed for skin necrosis, skin breakdown, infection. | 15 days

SECONDARY OUTCOMES:
The patients rated their pain experience by a visual analogue scale. The results were graded by Crawford's criteria. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Sumin Wen, M.D., Principal Investigator — The Second Hospital of Qinhuangdao
Locations (1):
- The second hospital of Qinhuangdao, Qinhuangdao, Hebei, China

REFERENCES:
- [Result] Lee YH, Kim JY, Chung MS, Baek GH, Gong HS, Lee SK. Two extension block Kirschner wire technique for mallet finger fractures. J Bone Joint Surg Br. 2009 Nov;91(11):1478-81. doi: 10.1302/0301-620X.91B11.22478. PMID 19880893